CLINICAL TRIAL: NCT05936216
Title: Expanded Access Use Of Tvi-Brain-1 For Treatment Of Recurrent Grade 4 Astrocytoma (Glioblastoma Multiforme; GBM)
Brief Title: TVI-Brain-1 in Expanded Access Patient
Status: No longer available | Type: Expanded Access
Sponsor: TVAX Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: TVI-AST-EAU
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Cancer Vaccines; Adjuvants, Immunologic

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: TVI-Brain 1 — Following surgery, tumor tissue is used to generate a cancer vaccine. Patients are vaccinated with neutralized cells to initiate an immune response. Following vaccinations, the patient's white blood cells are collected, the white blood cells are stimulated and expanded, and are then reinfused into the patient's blood.
  Other Names: Cancer vaccine plus immune adjuvant plus activated WBC

SUMMARY:
TVI-Brain-1 is being offered as a potential treatment option to a Named Patient (Emergency Use Authorization IND) for recurrent glioblastoma as there is no effective systemic treatment available for this disease or patient. TVI-Brain-1 is an experimental treatment that takes advantage of the fact that your body can produce immune cells, called 'killer' white blood cells that have the ability to kill large numbers of the cancer cells that are present in your body. TVI-Brain-1 is designed to generate large numbers of those 'killer' white blood cells and to deliver those cells into your body so that they can kill your cancer cells.

DETAILED DESCRIPTION:
The TVI-Brain-1 treatment involves several steps. First, the patient's cancer will be surgically removed to provide cells for the vaccine. Second, the patient will be vaccinated with the vaccine formulation. Third, the patient's blood will be filtered for killer T cell precursors which will then be cultured and stimulated to reach a higher (killer) activity level. Fourth, the activated cells will be infused into the patient's bloodstream so that they will be able to attack the cancer.

ELIGIBILITY:
Inclusion Criteria:

Recurrent glioblastoma diagnosis confirmed

* Age > 18
* Informed consent
* Diagnosis of grade IV glioma with progression following standard treatment.
* Must be able to tolerate surgery to provide tumor tissue for vaccine.
* Must be able to produce viable vaccine from tumor tissue.
* Karnofsky Performance Status must be 70 or greater.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Respiratory reserve must be reasonable.
* Sufficient renal function.
* Satisfactory blood counts.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Surgically removed cancer reveals that it is not grade IV glioma.
* Concomitant life-threatening disease.
* Active autoimmune disease.
* Currently receiving chemotherapy or biological therapy for the treatment of cancer.
* Currently receiving immunosuppressive drugs for any reason.
* Prior treatment with Avastin or other anti-angiogenesis treatment within 6 months.
* Prior treatment with Gliadel wafers.
* Corticosteroids beyond peri-operative period.
* Psychological, familial, sociological or geographical conditions that do not permit adequate medical follow-up and compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Providence St. Vincent Medical Center, Portland, Oregon, United States

REFERENCES:
- [Background] Sloan AE, Dansey R, Zamorano L, Barger G, Hamm C, Diaz F, Baynes R, Wood G. Adoptive immunotherapy in patients with recurrent malignant glioma: preliminary results of using autologous whole-tumor vaccine plus granulocyte-macrophage colony-stimulating factor and adoptive transfer of anti-CD3-activated lymphocytes. Neurosurg Focus. 2000 Dec 15;9(6):e9. doi: 10.3171/foc.2000.9.6.10. PMID 16817692
- [Background] Rosenberg SA, Packard BS, Aebersold PM, Solomon D, Topalian SL, Toy ST, Simon P, Lotze MT, Yang JC, Seipp CA, et al. Use of tumor-infiltrating lymphocytes and interleukin-2 in the immunotherapy of patients with metastatic melanoma. A preliminary report. N Engl J Med. 1988 Dec 22;319(25):1676-80. doi: 10.1056/NEJM198812223192527. PMID 3264384